CLINICAL TRIAL: NCT03694405
Title: A Randomized, Controlled Trial to Compare Protection in Adolescents Between Different Meningococcal Immunization Schedules Used in Canada; a Canadian Immunization Research Network (CIRN) Study.
Brief Title: Adolescent MenACWY Booster Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: University of British Columbia (Other); University of Calgary (Other); Canadian Center for Vaccinology (Other); Alberta Health services (Other); British Columbia Centre for Disease Control (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT17_CIRN24_Achieve01
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Meningococcal Disease, Invasive
Keywords: MenACWY; Neisseria meningitidis; adolescents
MeSH Terms: conditions — Meningococcal Infections | interventions — MenACWY-CRM vaccine; Meningococcal Vaccines; tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine

STUDY DESIGN:
Intervention Model Description: Group 1 = 3 prior doses of MenC vaccine (Alberta), Group 2 = 2 prior doses of MenC vaccine (British Columbia), Group 3 = 1 prior dose of MenC vaccine (Nova Scotia). Group A = Menveo (MenACWY-CRM), Group B = Menactra (MenACWY-DT), Group C = Nimenrix (MenACWY-TT)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Group 1A (Experimental): 3 doses prior MenC , randomized to receive MenACWY-CRM (Menveo)
  Interventions: Biological: MenACWY-CRM
- Group 1B (Experimental): 3 doses prior MenC, randomized to receive MenACWY-DT (Menactra)
  Interventions: Biological: MenACWY-DT
- Group 1C (Experimental): 3 doses prior MenC, randomized to receive MenACWY-TT (Nimenrix)
  Interventions: Biological: MenACWY-TT
- Group 2A (Experimental): 2 doses prior MenC, randomized to receive MenACWY-CRM (Menveo)
  Interventions: Biological: MenACWY-CRM
- Group 2B (Experimental): 2 doses prior MenC, randomized to receive MenACWY-DT (Menactra)
  Interventions: Biological: MenACWY-DT
- Group 2C (Experimental): 2 doses prior MenC, randomized to receive MenACWY-TT (Nimenrix)
  Interventions: Biological: MenACWY-TT
- Group 3A (Experimental): 1 dose prior MenC, randomized to receive MenACWY-CRM (Menveo)
  Interventions: Biological: MenACWY-CRM
- Group 3B (Experimental): 1 dose prior MenC, randomized to receive MenACWY-DT (Menactra)
  Interventions: Biological: MenACWY-DT
- Group 3C (Experimental): 1 dose prior MenC, randomized to receive MenACWY-TT (Nimenrix)
  Interventions: Biological: MenACWY-TT

INTERVENTIONS:
Biological: MenACWY-CRM — Booster vaccination with MenACWY-CRM
  Other Names: Menveo
  Arms: Group 1A; Group 2A; Group 3A
Biological: MenACWY-DT — Booster vaccination with MenACWY-DT
  Other Names: Menactra
  Arms: Group 1B; Group 2B; Group 3B
Biological: MenACWY-TT — Booster vaccination with MenACWY-TT
  Other Names: Nimenrix
  Arms: Group 1C; Group 2C; Group 3C

SUMMARY:
This study is to confirm non-inferiority of the three MenACWY vaccines (Menveo, Menactra or Nimenrix) in adolescents, and to identify whether the number of previous doses of MenC influences the response to the MenACWY vaccine.

DETAILED DESCRIPTION:
Participants will be randomized to receive one of the three doses of licensed MenACWY as a booster dose in adolescents. Serology will be collect at 3 time points; prior to the booster dose and 1 month and 1 year post-vaccination to measure antibody levels. The participants are healthy students in grades 7-9 who have not received their MenACWY vaccine yet and received their routine infant MenC vaccines per previous Canadian schedules.

ELIGIBILITY:
INCLUSION CRITERIA

All the following need to be fulfilled:

1. Healthy adolescent
2. Previous receipt of appropriate MenC vaccine according to the relevant provincial schedule (see above)
3. Parent/legal guardian has given informed consent OR participant has given consent (if participant demonstrates capacity to consent)
4. Participant has given consent (as above) OR assent.

EXCLUSION CRITERIA

The participant may not enter the trial if ANY of the following apply:

1. Has already received any doses of MenACWY vaccine at any age
2. Previous confirmed or suspected meningococcal disease
3. Close contact with an individual with laboratory-confirmed N. meningitidis in prior 12 months
4. Previous allergic reaction to a component of any of the 3 vaccines
5. Serious chronic or progressive disease
6. Confirmed/suspected immunodeficiency
7. Receipt of more than 1 week of immunosuppressants or immune modifying drugs (e.g. oral prednisolone >0.5mL/kg/day or intravenous glucocorticoid steroid). Nasal, topical or inhaled steroids are allowed
8. Administration of immunoglobulins within the prior 12 months and/or any blood products planned during the study period
9. Pregnancy (based on history from adolescent and parent/legal guardian)
10. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

TEMPORARY EXCLUSION CRITERIA If the adolescent has a temperature ≥ 38°C, then vaccination (and blood sampling if due to occur at same visit) will be postponed until resolution of fever.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Confirm non-inferiority of MenC protection at 1-year post-MenACWY booster between groups with differing priming schedules | 1 year following MenACWY adolescent booster
  N. meningitidis capsular group C serum bactericidal antibody titer
Confirm non-inferiority of MenC protection at 1-year post-MenACWY booster between differing vaccines | 1 year following MenACWY adolescent booster
  N. meningitidis capsular group C serum bactericidal antibody titer

SECONDARY OUTCOMES:
Confirm non-inferiority of MenC protection at 1 month post-MenACWY booster between groups with differing MenC priming schedules. | 1 month following MenACWY booster
  N. meningitidis capsular group C serum bactericidal antibody titer
Confirm non-inferiority of MenC protection at 1 month post-MenACWY booster between groups with different MenACWY vaccines | 1 month following MenACWY booster
  N. meningitidis capsular group C serum bactericidal antibody titer
Subgroup analysis to determine effects of different MenACWY vaccines in subjects primed with different MenC schedules at 1 month and 1 year post-MenACWY booster | 1 month and 1 year following MenACWY booster
  N. meningitidis capsular group C serum bactericidal antibody titer
Subgroup analysis to determine effects of different MenC priming schedules in subjects receiving different MenACWY booster immunizations at 1 month and 1 year post-MenACWY booster | 1 month and 1 year following MenACWY booster
  N. meningitidis capsular group C serum bactericidal antibody titer
Confirm safety of MenACWY conjugate vaccines | Up to 1 month post-vaccine
  Adverse events as reported by study participants

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sadarangani, BM BCh DPhil, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Children's Hospital Research Institute, University of Calgary, Calgary, Alberta
  - Vaccine Evaluation Center, BC Children's Hospital Research Institute, Vancouver, British Columbia
  - Canadian Center for Vaccinology, Halifax, Nova Scotia